CLINICAL TRIAL: NCT02841969
Title: Randomised Double Blind Controlled Trial of Neutral Electrolysed Water vs Conventional Management of Non-healing Diabetic Feet (NEWfeet)
Brief Title: Management of the Diabetic Foot Using Electrolysed Water
Acronym: NEWfeet
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Following consultation, neutral electrolysed water was deemed to be a medical device. A study amendment will re-submitted to NHS Ethics and the UK regulator (MHRA). These actions delayed due to the pandemic - expected to take place in June 2022.
Sponsor: NHS Lanarkshire (Other Government)
Collaborators: Aqualution Systems Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NEWfeet_01; L16077 (Other: NHS Lanarkshire)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Foot
Keywords: Ulcer; Electrolysed; Water
MeSH Terms: conditions — Diabetic Foot; Ulcer | interventions — superoxidized water

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal care - Prontosan (Active Comparator): Patient wounds will be irrigated using the in-use product (Prontosan)
  Interventions: Other: Prontosan
- Investigational arm - Electrolysed water (Experimental): Patient wounds will be irrigated using electrolysed water
  Interventions: Other: Electrolysed water

INTERVENTIONS:
Other: Electrolysed water — Irrigation of wound using electrolysed water
  Other Names: Aqualution Salvesan
  Arms: Investigational arm - Electrolysed water
Other: Prontosan — Irrigation of wound using Prontosan
  Arms: Normal care - Prontosan

SUMMARY:
More patients with diabetes mellitus have led to increasing rates of chronic non-healing wounds. These wounds are colonised with pathogens, including multi-drug resistant organisms. Despite repeated courses of antibiotics subsequent management is difficult due to devascularisation of surrounding tissues and healing failures. Ultimately, patients may require amputation. Electrolysed water is a novel antiseptic produced by passing an electric current through a mixture of tap water and salt. Microbiocidal activity is due to the presence of hypochlorous acid at neutral Ph. Irrigation of chronic wounds with electrolysed water reduces bacterial load and appears to encourage wound healing. Following an encouraging pilot study, we propose to compare electrolysed water against conventional management for diabetic patients with non-healing foot ulcers. Adult diabetics with chronic ulcers attending podiatry at Hairmyres Hospital will be recruited to receive regular debridement and irrigation of wounds using either in-use product (Prontosan™) or electrolysed water as part of a prospective randomised controlled trial. Strict enrolment criteria will be applied, with regular clinical assessment and microbiological screening. Lesions present for >6 weeks and >2cm will be photographed at trial entry and graded using standardised criteria. Wounds will be monitored for at least 12 weeks (max. 20), with primary composite end-point defined as complete healing; >50% healing of initial lesion; and/or avoidance of surgical intervention. Secondary endpoints are surgical intervention, including debridement or amputation; antibiotic therapy; and/or patient death. The main objective is to compare rapidity of wound healing using either in-use product or electrolysed water. Improved healing could potentially benefit patients who might otherwise progress to amputation. We will also monitor antimicrobial consumption in study patients throughout the trial. A final objective is to cost the use of electrolysed water vs cost of Prontosan in the routine management of diabetic foot ulcers.

DETAILED DESCRIPTION:
Study design: The entrance criteria specify adult diabetic patients (18-65 years) with chronic (>6 weeks) non-healing wounds(>2cm2) identified by study clinicians and counselled by aid of a Participant Information sheet (PIS). Having considered the PIS for >24hrs, patients who wish to participate will provide signed formal consent and will be entered into the trial. Relevant demographic and clinical data will be recorded with baseline microbiology, blood tests and classification of wound and pain score. Wounds will be graded according to the Texas classification and photographed. Pain score at entry will be measured by modified McGill questionnaire and graded from 0(no pain) to 5(severe pain). Study patients will be randomly assigned to receive either in-use product or electrolysed water according to predetermined statistical protocol and will be given a code for continued identification. The patient's notes will be tagged with study and code information, with copies sent to the patient's GP.

The wound will be inspected, debrided, cleaned and irrigated twice a week using electrolysed water or in-use product (Prontosan™). In-patients may receive more frequent application (e.g. daily) depending upon wound status. This will be performed by ward nurses for in-patients and for outpatients by podiatrists in the Diabetic clinic. Patients will be assessed by podiatrists weekly (<=20wks) or until an agreed end-point is reached; research assessments will coincide with routine outpatient clinic attendance or in-patient review to minimise patient inconvenience.

Release of electrolysed water will be coordinated by the research scientist. Supplies will be decanted into identical containers in order to blind staff as to product identity. The bottles will be labelled 'A' or 'B. Patients randomised to receive study or in-use irrigant will continue with the same product, to which they were initially assigned.

If a patient develops an infection, then they will receive clinical review and microbiological screening. These patients will continue with trial irrigants but will be offered appropriate antibiotics according to laboratory data. They will be encouraged to complete the trial but their data will be analysed separately on final analysis.

Patients with underlying terminal disease will be excluded from this trial along with patients with severe co-morbidities, e.g. morbidly obese; uncontrolled diabetes (HbA1c > 97 mmol/mol); gangrene; chronic leg oedema/venous disease; end-stage renal disease; untreatable ischaemic heart disease; HIV; etc. Patients with ongoing infection at trial entry will be treated and then reassessed. Any previous documented allergy to either Prontosan™ or electrolysed water will also necessitate exclusion. Any adverse effects thought to be due to either irrigant will prompt study withdrawal and investigation. If there is doubt over the continuation of the correctly assigned irrigant for a specific patient, then that patient's data will be labelled as such and noted for the final analysis. This will also be the case and/or if there are lapses of more than 4 treatment sessions during therapy. All data will be retained for the final project report.

The primary composite end-points are: complete healing; >50% healing of initial lesion; and/or avoidance of surgical intervention including amputation. Secondary endpoints are: surgical debridement including amputation; antibiotic consumption; and patient death. Each patient lesion will be photographed at the agreed end-point.

ELIGIBILITY:
Inclusion Criteria:

Adult diabetic patients (18-65 years) with chronic (>6 weeks) non-healing wounds(>2cm2) identified and counselled by study clinicians, along with additional information supplied by the Patient Information leaflet.

-

Exclusion Criteria:

Patients with underlying terminal disease will be excluded from this trial along with those with severe co-morbidities, e.g. morbidly obese; uncontrolled diabetes (HbA1c > 97 mmol/mol); gangrene; chronic leg oedema/venous disease; end-stage renal disease; untreatable ischaemic heart disease; HIV; etc. Patients with ongoing infection at trial entry will be treated and then reassessed. Any previous documented allergy to either Prontosan™ or electrolysed water will also exclude the patient. Any adverse effects thought to be due to either irrigant will necessitate study withdrawal and investigation. If there is doubt over the continuation of the correctly assigned irrigant for a specific patient, then that patient's data will be labelled as such and noted for the final analysis. This will also be the case and/or if there are lapses of more than 4 treatment sessions during therapy.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complete wound healing | 12 weeks
  Compare the use of neutral electrolysed water in the management of chronic diabetic foot ulcers against routine NHS management, which uses Prontosan for antiseptic irrigation.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Dancer (MBBS, FRCP), MD, Principal Investigator — NHS Lanarkshire
Locations (1):
- Hairmyres Hospital, East Kilbride, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No